CLINICAL TRIAL: NCT04962113
Title: Effect of Tub Bathing on Skin and Bilirubin Levels in Infants Undergoing Tunnel and LED of Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, SERAP ÖZDEMİR, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulUC-Pediatri
Record Dates: First submitted 2021-06-23; First posted 2021-07-14 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-05

CONDITIONS: Newborn Jaundice
Keywords: tube bath; skin care; phototherapy
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tunnel group Tube bath during the phototherapy (Experimental)
  Interventions: Other: TUBE BATH
- Tunnel group rutin care (No Intervention)
- LED group Tube bath during the phototherapy (Experimental)
  Interventions: Other: TUBE BATH
- LED group rutine care (No Intervention)

INTERVENTIONS:
Other: TUBE BATH — Wrap Tube Baht (immersion)
  Arms: LED group Tube bath during the phototherapy; Tunnel group Tube bath during the phototherapy

SUMMARY:
The study was conducted as a randomized controlled study to determine effect of tube bathing on skin and bilirubin levels in infants undergoing tunnel and LED of phototherapy. The population of the study consisted of term babies with the diagnosis of hyperbilirubinemia in Gaziantep Cengiz Gökçek Maternity and Pediatrics Hospital and Kilis State Hospital Neonatal Intensive Care Units (NICU) among November 2019-September 2020. The sample size was composed of a total of 140 babies, which were determined according to Power Analysis and met the case selection criteria. Accordingly, Thirty-five babies were randomly assigned to each group (Tunnel Group = experiment and control; LED Group = experiment and control). The babies in the experimental groups were given a tube bath at 6 and 12 hours after phototherapy started. On the other hand, the babies in the control groups were given routine cares in the units. Data were gathered 'Information and Registration Form', Neonatal Skin Risk Assessment Scale (NSRAS) and Neonatal Skin Condition Score (NSCS).

ELIGIBILITY:
Inclusion Criteria:

* The baby is receiving phototherapy due to physiological hyperbilirubinemia,
* Being a term newborn,
* Monitoring of the LED group in the incubator and the tunnel group in the tunnel phototherapy device,
* Parents' consent to participate in the study.

Exclusion Criteria:

* Rh incompatibility between mother and baby,
* Finding ABO non-compliance,
* Positive direct Coombs test,
* Presence of congenital anomaly or syndrome,
* Any surgical intervention has been or will be made,
* Having any skin lesions,
* The need for mechanical ventilation.

Ages: 0 Days to 1 Month | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Sample size | 1-2 month
  The sample size was composed of a total of 140 babies, which were determined according to Power Analysis and met the case selection criteria.
Divided groups | 1 month
  Thirty-five babies were randomly assigned to each group (Tunnel Group = experiment and control; LED Group = experiment and control).
Experiment difining and time | 12 month
  The babies in the experimental groups were given a tube bath at 6 and 12 hours after phototherapy started. On the other hand, the babies in the control groups were given routine cares in the units.
Measurement | First, 6-12-24 hours for each nerwborn
  Data were gathered 'Information and Registration Form', Neonatal Skin Risk Assessment Scale (NSRAS) and Neonatal Skin Condition Score (NSCS).
Biochemical measurement | First, 6-12-24 hours for each nerwborn
  Total serum bilirubin values obtained from patient files.
TSB Findings | 10 month
  When differences regarding decrease in 24-hour total serum bilirubin (TSB) levels were compared in all relevant experimental groups, statistically differences were observed (p˂ .001). In particular, the levels of bilirubin were listed as LED-trial, Tunnel-trial, Tunnel-control and LED-control, respectively. It is worthy to utter herein that the decline in TSB was more notable in bathing groups.
Skin care findings | 10 month
  Skin integrity and moisture balance were better in bathing groups than control groups, the best was in the Tunnel-experimental group and the worst was in the Tunnel-control group (p˂ .001).
Conclusion | 12 month
  Tube bath is suggested that decreasing total serum bilirubin level and maintaining skin integrity and moisture balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Serap ÖZDEMİR, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bagwell, G. A., & Steward, D. K. (2020). Hematologic System. Comprehensive Neonatal Nursing Care (6th ed.), Springer Publishing Company, 11C. New York, 315-335.
- [Background] Association of Women's Health, Obstetric and Neonatal Nurses. (2018). Evidence-Based Clinical Practice Guideline: Neonatal Skin Care (4th ed.). Washington, DC.
- [Background] Brogan J, Rapkin G. Implementing Evidence-Based Neonatal Skin Care With Parent-Performed, Delayed Immersion Baths. Nurs Womens Health. 2017 Dec;21(6):442-450. doi: 10.1016/j.nwh.2017.10.009. PMID 29223208
- [Background] Dağ, Y. S., & Yayan, E. H. (2019). The Effect on Bilirubin Levels of Massage, Tub Bath, and Sponge Bath in Newborns with Hyperbilirubinemia: A Randomized ControlLed Trial. European Journal of Integrative Medicine, 27, 70-74.
- [Background] Kaplan, M., Wong, RJ., Burgis, JC., Sibley E., Stevensen, DK. (2020). Neonatal Jaundice and Liver Diseases, Martin RJ, Fanoroff AA, Walsh MC, Fanaroff and Martin's Neonatal-Perinatal Medicine in 11th Edition, Philadelphia, 91:1788-1852.
- [Background] Mohammadi Pirkashani, L., Asghari, G., Marofi, M., & Barekatain, B. (2017). Effect of Chicory Extract Bath on Neonatal Bilirubin Levels: A Randomized Clinical Trial Study. International Journal of Pediatrics, 5(12), 6679-6688.
- [Background] Sherbiny HS, Youssef DM, Sherbini AS, El-Behedy R, Sherief LM. High-intensity light-emitting diode vs fluorescent tubes for intensive phototherapy in neonates. Paediatr Int Child Health. 2016 May;36(2):127-33. doi: 10.1179/2046905515Y.0000000006. PMID 25844870
- [Derived] Ozdemir S, Balci S. The Effect of Tub Bathing on the Skin and Bilirubin Levels of Babies Receiving Tunnel and Light-Emitting Diode Phototherapies: A Randomized Controlled Trial. Adv Skin Wound Care. 2024 Jul 1;37(7):1-9. doi: 10.1097/ASW.0000000000000163. PMID 38899824